CLINICAL TRIAL: NCT03899116
Title: Gradual Deflation of Thigh Tourniquet for Attenuation of Hemodynamic Post-tourniquet Response in Old Patients :Randomized Control Study
Brief Title: Gradual Deflation of Thigh Tourniquet for Attenuation of Hemodynamic Post-tourniquet Response in Old Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, Principal investigator, Cairo University
Other Study IDs: 101-2018
Record Dates: First submitted 2019-03-06; First posted 2019-04-02 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Tourniquet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- G50: The tourniquet cuff pressure will be deflated gradually by 50 mm Hg every 2 minutes till complete deflation.
  Interventions: Other: deflation of pneumatic tourniquet
- G100: The tourniquet cuff pressure will be deflated gradually by 100 mm Hg every 2 minutes till complete deflation.
  Interventions: Other: deflation of pneumatic tourniquet
- G0: The tourniquet cuff will be released till complete deflation.
  Interventions: Other: deflation of pneumatic tourniquet

INTERVENTIONS:
Other: deflation of pneumatic tourniquet — gradual deflation with variable degrees

SUMMARY:
Deflation of the pneumatic tourniquet used in lower limb surgery is usually associated with hemodynamic instability, metabolic and respiratory changes. These changes are usually tolerated by young, healthy patients; However, these complications are risky for elderly and cardiac patients. The aim of this study is to assess the effect of gradual deflation of thigh tourniquet on the hemodynamics and arterial blood gases compared to the usual practice

DETAILED DESCRIPTION:
Pneumatic tourniquet will be applied on the mid- thigh with cuff pressure of 350 mm Hg. After the end of surgery, the lower limb will be elevated at 45-degree and the patients will randomized into one of the three groups:

G 50 (n=30) : The tourniquet cuff pressure will be deflated gradually by 50 mm Hg every 2 minutes till complete deflation.

G 100 (n=30): The tourniquet cuff pressure will be deflated gradually by 100 mm Hg every 2 minutes till complete deflation.

G 0 (n=30): The tourniquet cuff will be released till complete deflation. If hypotension is observed during the procedure, it will be managed by 10 mg ephedrine.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective orthopedic lower limb surgery under pneumatic tourniquet

Exclusion Criteria:

* BMI ≥35Kg/ m2
* patients with unstable angina, left ventricular dysfunction , cerebrovascular disease ,bleeding disorders
* contraindication to tourniquet insertion
* patients requiring massive intraoperative blood transfusion (Blood loss more than 50% of the patients' blood volume (70 ml/Kg) ).

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients above 50 years scheduled for orthopedic lower limb surgery under pneumatic tourniquet
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
mean arterial blood pressure | 15 minutes after start of deflation of cuff
  The lowest mean arterial blood pressure during a 15-minute period after starting deflation of the tourniquet.

SECONDARY OUTCOMES:
hypotension | 15 minutes after start of deflation of cuff
  incidence of post tourniquet hypotension
cardiac output | 15 minutes after start of deflation of cuff
  cardiac output after starting deflation using non invasive electrical cardiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided